CLINICAL TRIAL: NCT02679560
Title: Effects of Liposomal Bupivacaine for Acute Pain in Hip and Femur Fractures: a Randomized, Active Comparator-controlled, Blinded Trial
Brief Title: Effects of Liposomal Bupivacaine for Acute Pain in Hip and Femur Fractures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Ian Elliott Brown (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ian Elliott Brown, Assistant Professor of Surgery, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 782382; D6.715L15J91110 (Other Grant/Funding Number: Defense Health Program)
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Femoral Fractures
Keywords: femur fracture, hip fracture, exparel, liposomal bupivacaine
MeSH Terms: conditions — Femoral Fractures; Hip Fractures | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): In patients with femur or hip fractures, a fascia iliaca compartment block using liposomal bupivacaine will be administered
  Interventions: Drug: Liposomal Bupivacaine
- Ropivacaine HCL (Placebo Comparator): In patients with femur or hip fractures, a fascia iliaca block using using 0.2% ropivacaine will be administered
  Interventions: Drug: Ropivacaine HCL

INTERVENTIONS:
Drug: Liposomal Bupivacaine — A fascia iliaca compartment block using liposomal bupivacaine will require less total opioid administration compared to a fascia iliaca block using 0.2% ropivacaine
  Other Names: Exparel®
  Arms: Liposomal Bupivacaine
Drug: Ropivacaine HCL — Ropivacaine HCL is a member of the amino amide class of local anesthetics. Naropin injection is a sterile, isotonic solution that contains the enantiomerically pure drug substance, sodium chloride for isotonicity and water for injection. It is administered parenterally.
  Other Names: Naropin (trade name)
  Arms: Ropivacaine HCL

SUMMARY:
This is an investigator-initiated, single-center, randomized, patient blinded, controlled trial. The purpose of this study is to compare the effect of a fascia iliaca compartment block (FICB) using 0.2% ropivacaine vs. liposomal bupivacaine in patients with femur and/or hip fractures admitted to the University of California Davis Medical Center (UCDMC). The primary endpoint will be the total opioid requirements during the 96 hour randomization period with secondary endpoints including total daily opioid requirements for days 1-4, duration of effect and objective pain scores using the numeric rating scale (NRS) during their hospital stay.

DETAILED DESCRIPTION:
In patients with femur or hip fractures, a fascia iliaca compartment block using liposomal bupivacaine will result in less total opioid administration during the randomization period compared to a fascia iliaca compartment block using 0.2% ropivacaine.

The long-term goal of this study is to provide pilot information to guide and design larger, multicenter trials which will evaluate the utility and cost-effectiveness of long acting liposomal bupivacaine as an opioid-sparring analgesic strategy in injured trauma patients. Ultimately, it is hoped that this information can improve safe and effective narcotic sparing analgesia in the awake, combat casualty, as well as serve as primary steps towards

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years ≤ 70 years
2. Patient's s/p trauma, with confirmed femur and/or hip fractures with a planned admission to the hospital
3. Patient is ambulatory without assistance (e.g. walker, cane, caretaker) prior to incident.

Exclusion Criteria:

1. >10 hours since presentation to the emergency department
2. History of seizure disorder, recent seizure or a document intra-cranial hemorrhage.
3. Central or peripheral neurologic deficit on presentation
4. Concern or compartment syndrome
5. Associated additional long bone fractures
6. End stage liver failure
7. Renal failure requiring dialysis
8. Pregnancy or breast feeding
9. Prisoners
10. Coagulopathy with INR >1.5
11. Use of direct thrombin inhibitors (bivalirudin, argatroban, desirudin, dabigatran etexilate), or direct factor Xa inhibitors (rivaroxaban, apixaban, edoxaban)
12. Suspected prolonged intubation within first 12 hours secondary to respiratory failure other than peri-procedurally
13. Adults unable to consent
14. Pediatric patients <18 years old
15. Patients exhibiting signs of shock upon admission, HR >120 or SBP <100 mmHg.
16. History of allergic reaction to local anesthetics
17. Administration of any other local anesthetic in the 2 hours prior to the study enrollment.
18. Distal femur fractures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Med Center- Trauma and Acute Care Surgery, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Ropivacaine HCL
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Ropivacaine HCL | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (0) | 33 (14) | 45 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Opioid Requirements
Description: Total opioid requirements during the 96 hour randomization period measured in milligram morphine equivalents
Time Frame: Assessment time frame will be the initial 96 hours of inpatient status after study drug administration with a daily assessment of total daily opioid requirements and objective pain scores using the numeric rating scale.
Population: There was a lack of enrollment and the sample size was too small to draw any results or conclusions for the study.
Arm/Group | Liposomal Bupivacaine | Ropivacaine HCL
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Outcomes
Description: Total daily opioid requirements for days 1-3, duration of effect and objective pain scores using the numeric rating scale (NRS) during their hospital stay
Time Frame: as for outcome 1
Population: There was a lack of enrollment and the sample size was too small to draw any results or conclusions for the study.
Arm/Group | Liposomal Bupivacaine | Ropivacaine HCL
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the participant's hospital stay up to 96 hours.
Arm/Group | Liposomal Bupivacaine | Ropivacaine HCL
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine (N=1) | Ropivacaine HCL (N=2)
Mild edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Mild edema at the site of IV placement.
mild muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hallucination (Psychiatric disorders) | 0 (0) | 1 (1) — one episode of nighttime hallucination
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — pruritus of lower extremity opposite injury
diaphoresis (Nervous system disorders) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
fever (Immune system disorders) | 0 (0) | 1 (1)
elevated systolic blood pressure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — present prior to study enrollment
tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — intermittent nausea post-op
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
moderate orthostatic hypotension (Nervous system disorders) | 0 (0) | 1 (1) — Moderate orthostatic hypotension (treated with normal saline bolus)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a lack of enrollment and the sample size was too small to draw any results or conclusions for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT02679560/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT02679560/ICF_001.pdf